CLINICAL TRIAL: NCT05211050
Title: Effect of Sumatriptan on Levcromakalim-Induced Symptoms in Individuals With Migraine: A Randomized Double-Blind Two-Way Crossover Study
Brief Title: Effect of Sumatriptan on Levcromakalim-Induced Symptoms in Individuals With Migraine
Acronym: SLIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Messoud Ashina, MD, Principal investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-21011542
Record Dates: First submitted 2022-01-04; First posted 2022-01-27 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Migraine Without Aura; Headache
MeSH Terms: conditions — Migraine without Aura; Headache | interventions — Cromakalim; Sumatriptan; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levcromakalim-Sumatriptan (Active Comparator): 20 participants with migraine without aura will receive a 20 min infusion of levcromakalim followed by a 10 min infusion of sumatriptan.
  Interventions: Drug: Levcromakalim; Drug: Sumatriptan
- Levcromakalim-Placebo (Placebo Comparator): 20 participants with migraine without aura will receive a 20 min infusion of levcromakalim followed by a 10 min infusion of saline.
  Interventions: Drug: Levcromakalim; Drug: Saline

INTERVENTIONS:
Drug: Levcromakalim — 20 min infusion of 1 mg Levcromakalim followed by either sumatriptan or placebo.
Drug: Sumatriptan — 10 min infusion of 4 mg sumatriptan.
  Arms: Levcromakalim-Sumatriptan
Drug: Saline — 10 min infusion of isotonic saline (placebo).
  Arms: Levcromakalim-Placebo

SUMMARY:
The study aims to explore the effects of Sumatriptan on Levcromakalim-induced migraine in individuals with migraine without aura.

DETAILED DESCRIPTION:
Opening of adenosine triphosphate-sensitive potassium (KATP) channels using Levcromakalim causes migraine attacks with and without aura in a high proportion of patients.

Sumatriptan has been shown to reverse Levcromakalim-induced dilation of the middle meningeal artery and headache in healthy volunteers, indicating that Sumatriptan can overturn the physiological effects of levcromakalim.

The study aims to explore the effects of Sumatriptan on Levcromakalim-induced migraine in individuals with migraine without aura.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided informed consent prior to initiation of any study-specific activities/procedures.
2. Age ≥18 years upon entry into screening.
3. History of migraine without aura for ≥12 months with a frequency of 1-5 migraine attacks per month before screening according to the International Headache Society (IHS) Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2018), based on medical records and/or patient self-report.

Exclusion Criteria:

1. History of any primary headache disorder other than migraine without aura, or tension-type headache with a frequency of ≥5 headache days per month before screening according to the International Headache Society (IHS) Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2018), based on medical records and/or patient self-report.
2. History of any secondary headache disorder before screening according to the International Headache Society (IHS) Classification ICHD-3 (Headache Classification Committee of the International Headache Society, 2018) based on medical records and/or patient self-report.
3. Any headache 48 hours prior to, or any migraine 72 hours prior to the start of the experiment on day 1 and 2.
4. Daily consumption of any drug/medication other than oral contraception (birth control).
5. Intake of prophylactic migraine medication within ≤30 days or 5 plasma half-lives (whichever is longer) prior to screening.
6. The participant is at risk of self-harm or harm to others as evidenced by past suicidal behavior.
7. History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the investigator will pose a risk to participant safety or interfere with the study evaluation, procedures or completion.
8. Female participants of childbearing potential with a positive pregnancy test assessed at screening or day 1 by a urine pregnancy test.
9. Female participants who are pregnant or breastfeeding or plan to become pregnant or breastfeed during participation in the study.
10. Evidence of current pregnancy or breastfeeding per participant self-report or medical records.
11. Participants likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures to the best of the participants' and investigator's knowledge.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
Incidence of migraine attacks | Assessed from baseline to 12 hours after infusion of levcromakalim.
  A migraine attack is defined as an attack fulfilling either (i) or (ii):
  (i) Headache fulfilling criteria C and D for migraine without aura according to the International Classification of Headache Disorders 3rd edition:
  C. Headache has at least two of the following characteristics:
  * unilateral location
  * pulsating quality
  * moderate or severe pain intensity (moderate to severe pain intensity is considered ≥4 on the numerical rating scale)
  * aggravation by cough (in-hospital phase) or causing avoidance of routine physical activity (out-hospital phase)
  D. During headache at least one of the following:
  * nausea and/or vomiting
  * photophobia and phonophobia
  (ii) Headache described as mimicking the patient's usual migraine attack and treated with acute migraine medication (rescue medication).

SECONDARY OUTCOMES:
Incidence of headache | Assessed from baseline to 12 hours after infusion of levcromakalim.
  Incidence of headache is defined as headache intensity ≥1 as measured by a numerical rating scale (NRS) from 0 to 10. It is a verbally declared scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Intensity of headache | Assessed from baseline to 12 hours after infusion of levcromakalim.
  Headache intensity scores are measured by a numerical rating scale (NRS). It is a verbally declared scale from 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Diameter of superficial temporal artery (STA) assessed using high frequency ultrasound | Assessed from baseline to 2 hours after infusion of levcromakalim.
  Diameter (mm) of superficial temporal artery (STA) is measured as a continuous outcome using high frequency ultrasound (Dermascan C, Cortex Technology, Denmark).
Incidence of adverse events | Assessed from baseline to 12 hours after infusion of levcromakalim.
  Participants are instructed to inform the investigators in the case of adverse events.

OTHER OUTCOMES:
Incidence of facial flushing | Assessed from baseline to 2 hours after infusion of levcromakalim.
  Incidence of facial skin flushing assessed by the investigator as a binary outcome.
Facial blood flow assessed using Laser Doppler Flowmetry | Assessed from baseline to 2 hours after infusion of levcromakalim.
  Facial blood flow is measured as a continuous outcome using Laser Doppler Flowmetry (LDI, Moor Instruments, Devon, United Kingdom).

CONTACTS AND LOCATIONS:
Overall Officials: Messoud Ashina, Prof., Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Centre, Glostrup, Region Sjælland, Denmark